CLINICAL TRIAL: NCT02366091
Title: Inflammation and Coronary Endothelial Function in Patients With Coronary Artery Disease
Brief Title: Inflammation and Coronary Endothelial Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: IRB00047206; R01HL120905 (NIH)
Record Dates: First submitted 2015-02-05; First posted 2015-02-19 (Estimated); Results first posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Methotrexate; Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Methotrexate (Experimental): Methotrexate 15 mg weekly by mouth and placebo for colchicine 1 tablet by mouth daily and folate 1 mg by mouth daily
  Interventions: Drug: Methotrexate; Drug: Placebo
- Colchicine (Experimental): Colchicine 0.6 mg daily by mouth and placebo for methotrexate 1 tablet weekly by mouth and folate 1 mg by mouth daily
  Interventions: Drug: Colchicine; Drug: Placebo
- Methotrexate & Colchicine (Experimental): Methotrexate 15 mg by mouth weekly and colchicine 0.6 mg by mouth daily and folate 1 mg by mouth daily
  Interventions: Drug: Methotrexate; Drug: Colchicine
- Placebo (Experimental): Placebo for methotrexate 1 tablet by mouth weekly and placebo for colchicine 1 tablet by mouth daily and folate 1 mg by mouth daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — Administered to determine the effect of anti-inflammatory agents on coronary and systemic endothelial function in patients with coronary artery disease
  Other Names: Trexall
  Arms: Methotrexate; Methotrexate & Colchicine
Drug: Colchicine — Administered to determine the effect of anti-inflammatory agents on coronary and systemic endothelial function in patients with coronary artery disease.
  Other Names: Colcrys
  Arms: Colchicine; Methotrexate & Colchicine
Drug: Placebo — Prepared by Johns Hopkins Investigational Drug Service to mimic methotrexate and colchicine.
  Other Names: A substance containing no medication
  Arms: Colchicine; Methotrexate; Placebo

SUMMARY:
The investigators are studying whether anti-inflammatory agents can improve abnormal coronary artery function in patients with coronary artery disease (CAD) and abnormal coronary artery endothelial function.

DETAILED DESCRIPTION:
Sometimes, in patients with coronary artery disease (CAD), even though blood pressure is controlled, the patients are on cholesterol medication, not smoking, eating properly and have normal levels of physical activity; the investigators still see development of new blockages, progression of existing blockages, and sometimes even clinical events like heart attacks and strokes. Therefore, the investigators are always trying to find additional ways to decrease the progression of existing blockages and to prevent new ones.

What the investigators are studying in this program is the function of the coronary arteries and in particular the inner lining of the arteries called the endothelium. It has several important functions; one of them is that under conditions of stress it releases a substance called nitric oxide which increases the size of the artery and increases blood flow. When it is not functioning normally the artery does not increase as much and blood flow does not increase during stress.

The investigators study coronary artery function with magnetic resonance imaging, or MRI. MRI is a method of obtaining images of what is happening inside the body. MRI does not involve radiation, x-ray, and injection of contrast. The investigators can measure flow in the artery and the dimension of the artery at rest and with a handgrip stress and learn the extent to which the artery dilates and flow increases with the stress. The investigators believe that inflammation can interfere with normal function and that by decreasing inflammation abnormal endothelial function may be improved.

Methotrexate and colchicine are anti-inflammatory agents approved by the Food and Drug Administration (FDA) to treat arthritis and some other conditions. These drugs are not approved for use to suppress inflammation in patients with coronary artery disease and improve coronary artery endothelial function. The FDA is allowing the use of methotrexate, colchicine and/or their combination in this research study.

This study will involve 24 weeks of anti-inflammatory drugs and 3 Magnetic Resonance Imaging (MRI) scans of the heart and other study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Participants of either gender who are 21 years of age (no upper age limit),
* History of prior Myocardial Infarction (MI), coronary revascularization, or coronary angiography or Multidetector Computer Tomography (MDCT) demonstrating at least one coronary artery with >50% luminal stenosis and no plans for revascularization,
* Clinically stable for 3 months,
* Vascular inflammation based on elevated hsCRP (>2mg L-1), or a clinical diagnosis of diabetes mellitus or metabolic syndrome (metabolic syndrome is defined by three or more of the following): Abdominal obesity (waist circumference: Men>102 cm (>40 in), Women >88 cm (>35 in)), Serum triglycerides ≥150 mg/dL (or taking medication to treat high triglycerides), HDL cholesterol: Men<40 mg/dL, Women<50 mg/dL (or taking medication to treat low HDL cholesterol), High blood pressure: ≥130/≥85 mm Hg (or taking medication to treat high blood pressure), or Fasting glucose: ≥100 mg/dL (or taking medication to treat high fasting glucose).
* Abnormal Coronary Endothelial Function (CEF) (change in CSA during IHE of <0% of the resting value: by this we mean any decrease in CSA or no change (0%) from baseline during IHE),
* Permission of patient's clinical attending physician,
* Patients being treated with a statin.

Exclusion Criteria:

* Patients unable to understand the risks, benefits, and alternatives of participation and give meaningful consent,
* Patients with contraindications to MRI such as implanted metallic objects (pre-existing cardiac pacemakers, cerebral clips) or indwelling metallic projectiles,
* Acute coronary syndrome within the prior three months,
* Pregnant women,
* Contraindications to methotrexate or colchicine as outlined by the American College of Rheumatology; including active bacterial infection, tuberculosis, or herpes zoster infection, leukopenia (<4000/mm3), thrombocytopenia (<135,000/mm3), elevation in hepatic transaminases (>2x upper limit of normal), hepatitis B or C, moderate renal disease (estimated creatine clearance <45ml/min), or planned surgery,
* Chronic inflammatory condition such as lupus or rheumatoid arthritis, ulcerative colitis or Crohn's disease,
* Interstitial lung disease or pulmonary fibrosis,
* HIV positive,
* Requirement for, or intolerance to, methotrexate or colchicine ,
* Intolerance to methotrexate, colchicine or folate,
* History of non-basal cell malignancy or treatment for lymphoproliferative disease in the past 5 years,
* Requirement for use of drugs that alter folate metabolism,
* History of alcohol abuse or unwillingness to limit consumption to < 4 drinks per week,
* Women of childbearing potential or intention to breastfeed.
* Men who plan to father children during the study period; men who have sexual intercourse with women of childbearing potential must agree to use a condom,
* Chronic use of oral or IV steroid therapy or other immunosuppressive or biologic response modifiers,
* History of chronic pericardial effusion, pleural effusion or ascites,
* New York Heart Association Class IV heart failure.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Weiss, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Everett BM, Pradhan AD, Solomon DH, Paynter N, Macfadyen J, Zaharris E, Gupta M, Clearfield M, Libby P, Hasan AA, Glynn RJ, Ridker PM. Rationale and design of the Cardiovascular Inflammation Reduction Trial: a test of the inflammatory hypothesis of atherothrombosis. Am Heart J. 2013 Aug;166(2):199-207.e15. doi: 10.1016/j.ahj.2013.03.018. Epub 2013 May 3. PMID 23895801
- [Background] Nidorf SM, Eikelboom JW, Budgeon CA, Thompson PL. Low-dose colchicine for secondary prevention of cardiovascular disease. J Am Coll Cardiol. 2013 Jan 29;61(4):404-410. doi: 10.1016/j.jacc.2012.10.027. Epub 2012 Dec 19. PMID 23265346
- [Background] Hays AG, Hirsch GA, Kelle S, Gerstenblith G, Weiss RG, Stuber M. Noninvasive visualization of coronary artery endothelial function in healthy subjects and in patients with coronary artery disease. J Am Coll Cardiol. 2010 Nov 9;56(20):1657-65. doi: 10.1016/j.jacc.2010.06.036. PMID 21050976
- [Background] Hays AG, Stuber M, Hirsch GA, Yu J, Schar M, Weiss RG, Gerstenblith G, Kelle S. Non-invasive detection of coronary endothelial response to sequential handgrip exercise in coronary artery disease patients and healthy adults. PLoS One. 2013;8(3):e58047. doi: 10.1371/journal.pone.0058047. Epub 2013 Mar 11. PMID 23536782
- [Background] Hays AG, Kelle S, Hirsch GA, Soleimanifard S, Yu J, Agarwal HK, Gerstenblith G, Schar M, Stuber M, Weiss RG. Regional coronary endothelial function is closely related to local early coronary atherosclerosis in patients with mild coronary artery disease: pilot study. Circ Cardiovasc Imaging. 2012 May 1;5(3):341-8. doi: 10.1161/CIRCIMAGING.111.969691. Epub 2012 Apr 5. PMID 22492483
- [Background] Weiss RG, Bottomley PA, Hardy CJ, Gerstenblith G. Regional myocardial metabolism of high-energy phosphates during isometric exercise in patients with coronary artery disease. N Engl J Med. 1990 Dec 6;323(23):1593-600. doi: 10.1056/NEJM199012063232304. PMID 2233948
- [Derived] Hays AG, Schar M, Bonanno G, Lai S, Meyer J, Afework Y, Steinberg A, Stradley S, Gerstenblith G, Weiss RG. Randomized Trial of Anti-inflammatory Medications and Coronary Endothelial Dysfunction in Patients With Stable Coronary Disease. Front Cardiovasc Med. 2021 Oct 15;8:728654. doi: 10.3389/fcvm.2021.728654. eCollection 2021. PMID 34722661

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 enrolled participants were excluded from the study prior to randomization as follows: 9 did not qualify by screening MRI; 3 did not qualify by lab work; 3 declined to proceed after qualifying by MRI; 2 were not randomized as enrollment target was met.
Period: Overall Study
Arm/Group | Methotrexate | Colchicine | Methotrexate & Colchicine | Placebo
Started | 24 | 23 | 24 | 23
Completed | 21 | 16 | 21 | 22
Not Completed | 3 | 7 | 3 | 1
Not completed — Withdrawal by Subject | 3 | 7 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Colchicine | Methotrexate & Colchicine | Placebo | Total
Number analyzed (Participants) | 24 | 23 | 24 | 23 | 94
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 61.6 [56.7 to 68.7] | 66.8 [56.2 to 67.9] | 63.4 [56.9 to 70.7] | 63.9 [55.9 to 69.5] | 63.77 [56.23 to 69.02]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 3 | 2 | 13
  Male | 18 | 21 | 21 | 21 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 23 | 22 | 23 | 22 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 2 | 2 | 9
  White | 20 | 19 | 21 | 19 | 79
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Coronary Cross Sectional Area (CSA) From Rest to That During Isometric Handgrip Exercise (IHE)
Description: Coronary segment endothelial function, measured by MRI as the percent change in coronary cross sectional area (CSA) from rest to that during isometric handgrip exercise (IHE) (as % rest) at 8 weeks.
Time Frame: At 8 weeks
Measure: Mean (Standard Error); unit: Percent change from rest measurement
Arm/Group | Methotrexate | Colchicine | Methotrexate & Colchicine | Placebo
Number analyzed (Participants) | 21 | 16 | 21 | 22
Percent change from rest measurement | -1.70 (2.85) | 2.71 (3.74) | -0.39 (2.23) | 2.04 (2.05)

2. Secondary Outcome: Percent Change in Coronary Cross Sectional Area (CSA) From Rest to That During Isometric Handgrip Exercise (IHE)
Description: Change in coronary segment endothelial function, measured by MRI as the percent change in coronary cross sectional area (CSA) from rest to that during isometric handgrip exercise (IHE) (as % rest) at 24 weeks.
Time Frame: At 24 weeks
Population: Not all participants who completed the primary outcome at 8 weeks went on to complete the 24 week studies, resulting in different numbers of participants analyzed between weeks 8 and 24.
Measure: Mean (Standard Error); unit: Percent change from rest measurement
Arm/Group | Methotrexate | Colchicine | Methotrexate & Colchicine | Placebo
Number analyzed (Participants) | 18 | 12 | 17 | 20
Percent change from rest measurement | 1.94 (3.36) | -5.39 (3.91) | 2.64 (2.60) | 9.26 (2.91)

3. Secondary Outcome: Percent Change in Coronary Blood Flow (CBF), Measured by MRI as the Change From Rest to IHE Stress
Description: Change in coronary blood flow (CBF), measured by MRI as the percent change from rest to IHE stress (as % rest) at 8 weeks.
Time Frame: At 8 weeks
Measure: Mean (Standard Error); unit: Percent change from rest measurement
Arm/Group | Methotrexate | Colchicine | Methotrexate & Colchicine | Placebo
Number analyzed (Participants) | 21 | 16 | 21 | 22
Percent change from rest measurement | 10.23 (4.70) | 14.06 (4.57) | 12.38 (5.58) | 13.81 (4.68)

4. Secondary Outcome: Serum High-sensitivity C Reactive Protein (Hs-CRP)
Description: Serum high-sensitivity C reactive protein (hs-CRP), measured by laboratory assessment in mg/l at 8 weeks.
Time Frame: At 8 weeks
Measure: Mean (Standard Error); unit: mg/l
Arm/Group | Methotrexate | Colchicine | Methotrexate & Colchicine | Placebo
Number analyzed (Participants) | 21 | 16 | 21 | 22
mg/l | 2.40 (0.54) | 3.10 (1.68) | 1.45 (0.22) | 1.65 (0.39)

5. Secondary Outcome: Serum Interleukin-6 (IL-6)
Description: Serum interleukin-6 (IL-6), measured by laboratory assessment in pg/ml at 8 weeks.
Time Frame: At 8 weeks
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Methotrexate | Colchicine | Methotrexate & Colchicine | Placebo
Number analyzed (Participants) | 21 | 16 | 21 | 22
pg/ml | 1.61 (0.55) | 1.20 (0.27) | 0.83 (0.07) | 0.92 (0.07)

6. Secondary Outcome: Brachial Flow Mediated Dilation (FMD)
Description: Brachial flow mediated dilation (FMD), measured as percent brachial artery dilation by ultrasound at 8 weeks.
Time Frame: At 8 weeks
Measure: Mean (Standard Error); unit: percent brachial artery dilation
Arm/Group | Methotrexate | Colchicine | Methotrexate & Colchicine | Placebo
Number analyzed (Participants) | 21 | 16 | 21 | 22
percent brachial artery dilation | 4.37 (0.70) | 3.23 (0.52) | 3.58 (0.48) | 4.57 (0.60)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over study enrollment and up to 4 weeks after the last dose of the study drug (total up to 28 weeks after initiation of study drug).
Arm/Group | Methotrexate | Colchicine | Methotrexate & Colchicine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 3/24 | 2/23 | 0/24 | 1/23
Other Adverse Events (participants affected / at risk) | 22/24 | 21/23 | 23/24 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate (N=24) | Colchicine (N=23) | Methotrexate & Colchicine (N=24) | Placebo (N=23)
Hospitalization (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Hospitalization for unstable angina/chest pain
Hospitalization (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Hospitalization for shoulder pain
Hopsitalization (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization for transient bilateral vision loss.
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hospitalization for pulmonary symptoms
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate (N=24) | Colchicine (N=23) | Methotrexate & Colchicine (N=24) | Placebo (N=23)
Infection (Infections and infestations) | 8 (8) | 8 (8) | 9 (9) | 6 (6)
Gastrointestinal disorder (Gastrointestinal disorders) | 9 (9) | 9 (9) | 7 (7) | 2 (2)
Joint/Muscle Soreness/Stiffness (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 7 (7) | 7 (7)
Chest Pain (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Extremity swelling (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Dental pain/infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Physical Injury (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 1 (1) | 2 (2)
Anxiety/Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Increased Alanine Amino Trans (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased White Blood Cell (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Decreased Hematocrit (Blood and lymphatic system disorders) | 4 (4) | 6 (6) | 8 (8) | 6 (6)
Decreased Estimated GFR (Renal and urinary disorders) | 5 (5) | 1 (1) | 3 (3) | 4 (4)
Increased Aspartate Amino Trans >3 x the normal range (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT02366091/Prot_SAP_000.pdf